CLINICAL TRIAL: NCT02257736
Title: A Phase 3 Randomized, Placebo-controlled Double-blind Study of JNJ-56021927 in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Subjects With Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: An Efficacy and Safety Study of Apalutamide (JNJ-56021927) in Combination With Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Participants With Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR105505; 56021927PCR3001 (Other: Janssen Research & Development, LLC); 2014-001718-25 (EudraCT Number); 2023-508606-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; JN56021927; ZYTIGA; Prednisone; Abiraterone acetate; Apalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Group 1: AAP and apalutamide (Experimental): Participants will receive apalutamide 240 milligram (mg) (4*60 mg tablets) and abiraterone acetate (AA) 1000 mg (4*250 mg tablets) once daily on an empty stomach and 5 mg prednisone (P), AAP, twice daily, until disease progression, unacceptable toxicity or end of treatment, whichever occurs first. After unblinding participants will be offered further treatment as defined in the Open-Label Extension (OLE) or Long-Term Extension (LTE) phase (AAP + open label apalutamide or AAP alone).
  Interventions: Drug: Apalutamide; Drug: Abiraterone acetate; Drug: Prednisone
- Group 2: AAP and Placebo (Placebo Comparator): Participants will receive matching Placebo of apalutamide and abiraterone acetate (AA) 1000 mg (4*250 mg tablets) once daily on an empty stomach and 5 mg prednisone (P), AAP, twice daily until disease progression, unacceptable toxicity or end of treatment, whichever occurs first. After unblinding participants will be offered further treatment as defined in the OLE or LTE phase (AAP + open label apalutamide or AAP alone).
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Apalutamide — Participants will receive 240 mg (4*60 mg tablets) of apalutamide once daily orally.
  Arms: Group 1: AAP and apalutamide
Drug: Abiraterone acetate — Participants will receive 1000 mg (4*250 mg tablets) of abiraterone acetate (AA) once daily orally.
  Other Names: ZYTIGA
Drug: Prednisone — Participants will receive 5 mg tablet of prednisone twice daily orally.
Drug: Placebo — Participants will receive matching placebo to apalutamide once daily orally.
  Arms: Group 2: AAP and Placebo

SUMMARY:
The purpose of this study is to compare the radiographic progression-free survival (rPFS) of apalutamide in combination with abiraterone acetate (AA) plus prednisone or prednisolone (AAP) and AAP in participants with chemotherapy-naive (participants who did not receive any chemotherapy [treatment of cancer using drugs]) metastatic castration-resistant prostate cancer (mCRPC) (cancer of prostate gland [gland that makes fluid that aids movement of sperm]).

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither the Investigator nor the participant know the treatment) placebo-controlled and multicenter (when more than 1 hospital or medical school team work on a medical research study) study to determine if participants with chemotherapy-naive mCRPC will benefit from the addition of apalutamide to AAP compared with AAP alone. The study consists of 3 phases: Screening phase; Treatment phase, and Follow-up phase. At the final analysis, the study will be unblinded. After the Independent Data Monitoring Committee (IDMC) review and the sponsor's subsequent decision participants will be offered to receive treatment either in the Open-Label Extension Phase or the Long-Term Extension Phase of study. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate
* Metastatic disease as documented by technetium-99m (99mTc) bone scan or metastatic lesions by computed tomography (CT) or magnetic resonance imaging (MRI) scans (visceral or lymph node disease). If lymph node metastasis is the only evidence of metastasis, it must be greater than or equal to (>=) 2 centimeter (cm) in the longest diameter
* Castration-resistant prostate cancer demonstrated during continuous androgen deprivation therapy (ADT), defined as 3 rises of PSA, at least 1 week apart with the last androgen deprivation therapy (PSA) >= 2 nanogram per milliliters (ng/mL)
* Participants who received a first generation anti-androgen (eg, bicalutamide, flutamide, nilutamide) must have at least a 6-week washout prior to randomization and must show continuing disease (PSA) progression (an increase in PSA) after the washout period
* Prostate cancer progression documented by prostate-specific antigen (PSA) according to the Prostate Cancer Clinical Trials Working Group (PCWG2) or radiographic progression of soft tissue according to modified Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST) modified based on PCWG2, or radiographic progression of bone according to PCWG2
* Participants who cross-over from Prednisone alone to open-label apalutamide plus AAP should still be in the double-blind phase of the study, should be receiving AAP alone and should have ECOG 0-1-2.

Exclusion Criteria:

* Small cell or neuroendocrine carcinoma of the prostate
* Known brain metastases
* Prior chemotherapy for prostate cancer, except if administered in the adjuvant/neoadjuvant setting
* Previously treated with ketoconazole for prostate cancer for greater than 7 days
* Therapies that must be discontinued or substituted at least 4 weeks prior to randomization include the following: a) Medications known to lower the seizure threshold, b) Herbal and non-herbal products that may decrease PSA levels (example [eg], saw palmetto, pomegranate) or c) Any investigational agent
* At Screening need for parenteral or oral opioid analgesics (eg, codeine, dextropropoxyphene)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (173):
- United States (46):
  - Phoenix, Arizona
  - La Mesa, California
  - Los Angeles, California
  - Modesto, California
  - San Diego, California
  - San Francisco, California
  - Santa Barbara, California
  - Aurora, Colorado
  - Denver, Colorado
  - Jensen Beach, Florida
  - Lakeland, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Atlanta, Georgia
  - Melrose, Illinois
  - Niles, Illinois
  - Marrero, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Auburn, Maine
  - Baltimore, Maryland
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Albany, New York
  - Johnson City, New York
  - New York, New York
  - Poughkeepsie, New York
  - Syracuse, New York
  - The Bronx, New York
  - Columbus, Ohio
  - Tualatin, Oregon
  - Lancaster, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Auburn, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Wenatchee, Washington
  - Madison, Wisconsin
- Argentina (6):
  - Ciudad Automoma Buenos Aires
  - Ciudad de Buenos Aires
  - Córdoba
  - La Rioja
  - Mendoza
  - Rosario
- Australia (11):
  - Adelaide
  - Ashford
  - Camperdown
  - Herston
  - Liverpool
  - Malvern
  - Melbourne
  - Southport
  - Wahroonga
  - West Heidelberg
  - Woolloongabba
- Belgium (10):
  - Antwerp
  - Brussels
  - Ghent
  - Gosselies
  - Leuven
  - Liège
  - Namur
  - Ottignies
  - Roeselare
  - Sint-Niklaas
- Brazil (6):
  - Barretos
  - Ijuí
  - Natal
  - Porto Alegre
  - São José do Rio Preto
  - São Paulo
- Canada (12):
  - Abbotsford, British Columbia
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - London, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Weston, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- France (9):
  - Angers
  - Caen
  - Dijon
  - Le Mans
  - Lyon
  - Montpellier
  - Paris
  - Saint-Herblain
  - Toulouse
- Germany (8):
  - Berlin
  - Dresden
  - Freiburg im Breisgau
  - Hamburg
  - Heidelberg
  - Münster
  - Nürtingen
  - Wuppertal
- Japan (15):
  - Fukuoka
  - Kanazawa
  - Kashiwa
  - Kita-Gun
  - Kumamoto
  - Kurume
  - Matsuyama
  - Miyazaki
  - Nagasaki
  - Osaka
  - Ōsaka-sayama
  - Sakura
  - Sapporo
  - Ube
  - Yokohama
- Mexico (6):
  - Chihuahua City
  - Cuernavaca
  - Culiacán
  - México
  - Oaxaca City
  - Zapopan
- Netherlands (10):
  - Amsterdam
  - Amsterdam-Zuidoost
  - Blaricum
  - Dordrecht
  - Groningen
  - Heerlen
  - Nieuwegein
  - Nijmegen
  - Rotterdam
  - The Hague
- Russia (7):
  - Kursk
  - Moscow
  - Omsk
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Ufa
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Pretoria
- South Korea (3):
  - Goyang-si
  - Seongnam
  - Seoul
- Spain (7):
  - Alcorcón
  - Barcelona
  - Cadiz
  - Córdoba
  - Madrid
  - San Sebastián de los Reyes
  - Valencia
- United Kingdom (13):
  - Ayr
  - Belfast
  - Birmingham
  - Edinburgh
  - Glasgow
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Plymouth
  - Preston
  - Stevenage
  - Sutton
  - Westcliff-on-Sea

REFERENCES:
- [Derived] Roy S, Wallis CJD, Morgan SC, Kishan AU, Le ATT, Malone J, Sun Y, Spratt DE, Saad F, Malone S. Implications of metastatic stage at presentation in docetaxel naive metastatic castrate resistant prostate cancer. Prostate. 2023 Jul;83(10):912-921. doi: 10.1002/pros.24512. Epub 2023 Apr 18. PMID 37071764
- [Derived] Saad F, Efstathiou E, Attard G, Flaig TW, Franke F, Goodman OB Jr, Oudard S, Steuber T, Suzuki H, Wu D, Yeruva K, De Porre P, Brookman-May S, Li S, Li J, Thomas S, Bevans KB, Mundle SD, McCarthy SA, Rathkopf DE; ACIS Investigators. Apalutamide plus abiraterone acetate and prednisone versus placebo plus abiraterone and prednisone in metastatic, castration-resistant prostate cancer (ACIS): a randomised, placebo-controlled, double-blind, multinational, phase 3 study. Lancet Oncol. 2021 Nov;22(11):1541-1559. doi: 10.1016/S1470-2045(21)00402-2. Epub 2021 Sep 30. PMID 34600602

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment disposition has been reported in participant flow.
Groups:
- Placebo+ Abiraterone Acetate - Prednisolone: Participants received 4*60 milligrams (mg) tablets of matching placebo orally once daily (qd) with or without food and 4*250 mg tablets of abiraterone acetate (AA) orally qd on empty stomach followed by prednisolone 5 mg orally twice daily with food for 24 cycles (each cycle was equal to 28 days), and thereafter every 3 cycles. Participants received treatment until radiographic progression or unequivocal clinical progression, unacceptable toxicity, or death.
- Apalutamide + Abiraterone Acetate - Prednisolone: Participants received 4*60 mg tablets of apalutamide tablets orally qd with or without food and 4*250 mg tablets of AA orally qd on empty stomach followed by prednisolone 5 mg orally twice daily with food for 24 cycles, and thereafter every 3 cycles. Participants received treatment until radiographic progression or unequivocal clinical progression, unacceptable toxicity, or death.
Period: Overall Study
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Started | 490 | 492
Completed | 39 | 45
Not Completed | 451 | 447
Not completed — Progressive disease | 365 | 327
Not completed — Adverse Event | 45 | 56
Not completed — Withdrawal by Subject | 21 | 38
Not completed — Death | 11 | 6
Not completed — Physician Decision | 5 | 9
Not completed — Non-Compliance with study drug | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 7
Not completed — Randomized, not treated | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone | Total
Number analyzed (Participants) | 490 | 492 | 982
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (8.06) | 71.4 (8.34) | 71.1 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 490 | 492 | 982
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 50 | 104
  Not Hispanic or Latino | 411 | 422 | 833
  Unknown or Not Reported | 25 | 20 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 9 | 17
  Asian | 53 | 58 | 111
  Black or African American | 18 | 19 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 373 | 365 | 738
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 40
  Other | 18 | 21 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 3 | 3 | 6
  AUSTRALIA | 31 | 47 | 78
  BELGIUM | 16 | 16 | 32
  BRAZIL | 21 | 18 | 39
  CANADA | 12 | 18 | 30
  FRANCE | 18 | 16 | 34
  GERMANY | 10 | 9 | 19
  ITALY | 33 | 36 | 69
  JAPAN | 23 | 27 | 50
  MEXICO | 19 | 16 | 35
  NETHERLANDS | 14 | 16 | 30
  RUSSIAN FEDERATION | 59 | 46 | 105
  SOUTH AFRICA | 9 | 8 | 17
  SOUTH KOREA | 28 | 29 | 57
  SPAIN | 43 | 36 | 79
  UNITED KINGDOM | 23 | 27 | 50
  UNITED STATES | 128 | 124 | 252

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: The rPFS was defined as the time from randomization to the occurrence of one of the following: 1) a participant was considered to have progressed by bone scan if - a) the first bone scan with greater than or equal to (>=) 2 new lesions compared to baseline was observed in less than (<) 12 weeks from randomization and was confirmed by a second bone scan taken >=6 weeks later showing >=2 additional new lesions (a total of >=4 new lesions compared to baseline), b) the first bone scan with >=2 new lesions compared to baseline was observed in >=12 weeks from randomization and the new lesions were verified on the next bone scan >=6 weeks later (a total of >=2 new lesions compared to baseline); 2) progression of soft tissue lesions measured by computerized tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Time Frame: Up to 3 years and 4 months
Population: Intent-to-treat (ITT) population included all randomized participants who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Number analyzed (Participants) | 490 | 492
months | 16.59 [13.86 to 19.32] | 23.98 [19.71 to 27.50]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS was defined as the time from randomization to date of death from any cause.
Time Frame: Up to 5 years and 10 months
Population: ITT population included all randomized participants who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Number analyzed (Participants) | 490 | 492
months | 33.71 [31.24 to 38.28] | 36.17 [32.76 to 38.77]

3. Secondary Outcome: Time to Chronic Opioid Use
Description: Time to chronic opioid use was defined as the time from date of randomization to the first date of opioid use.
Time Frame: Up to 5 years and 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Number analyzed (Participants) | 490 | 492
months | 53.26 [42.02 to NA] — Here 'NA' represents that upper limit of CI was not estimable due to lesser number of events. | 46.98 [39.23 to NA] — Here 'NA' represents that upper limit of CI was not estimable due to lesser number of events.

4. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: Time to initiation of cytotoxic chemotherapy was defined as the time from date of randomization to the date of initiation of cytotoxic chemotherapy.
Time Frame: Up to 5 years and 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Number analyzed (Participants) | 490 | 492
months | 34.23 [29.54 to 39.16] | 36.11 [32.23 to 42.55]

5. Secondary Outcome: Time to Pain Progression
Description: Time to pain progression: time from randomization to first date that participant either experienced an increase by 2 points from baseline in Brief Pain Inventory Short Form (BPI-SF) worst pain intensity item (item 3) or Case Report Form (CRF) pain, observed at 2 consecutive evaluations >=4 wks apart, or initiation of chronic opioids as defined in time to chronic opioid use, whichever occurred first. BPI-SF is a self-administered questionnaire developed to assess severity of pain and impact of pain on daily functions. Item 3(worst pain intensity) asks participants to rate worst pain in prior 7-days on a 0-10 numeric rating scale, where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine." A lower score is better.CRF pain refers to participant's response to global pain assessment "How would you rate your pain over the past 7 days?"with a scale of 0("No pain") to 10("Pain as bad as you can imagine"),that is systematically reported and recorded on the eCRF.
Time Frame: Up to 5 years and 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
Number analyzed (Participants) | 490 | 492
months | 26.51 [22.57 to 29.50] | 21.82 [17.97 to 25.66]

ADVERSE EVENTS:
Time Frame: Up to 3 years and 4 months
Description: Safety Analysis set included all participants who received at least 1 dose of study drug, with treatment assignments designated according to actual study treatment received.
Arm/Group | Placebo+ Abiraterone Acetate - Prednisolone | Apalutamide + Abiraterone Acetate - Prednisolone
All-Cause Mortality (participants affected / at risk) | 350/489 | 338/490
Serious Adverse Events (participants affected / at risk) | 166/489 | 192/490
Other Adverse Events (participants affected / at risk) | 459/489 | 472/490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ Abiraterone Acetate - Prednisolone (N=489) | Apalutamide + Abiraterone Acetate - Prednisolone (N=490)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 4 | 4
Angina Pectoris (Cardiac disorders) | 0 | 4
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 6 | 3
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac Failure (Cardiac disorders) | 3 | 2
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 4 | 4
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 6
Palpitations (Cardiac disorders) | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0
Stress Cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 2
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Diplopia (Eye disorders) | 1 | 0
Visual Impairment (Eye disorders) | 0 | 1
Anal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 2 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 3
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0
Lumbar Hernia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Periodontal Disease (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 5 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 2 | 4
Fatigue (General disorders) | 0 | 1
Gait Inability (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 3 | 0
Generalised Oedema (General disorders) | 1 | 0
Granuloma (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 3 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 5
Oedema Peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 2
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Contrast Media Allergy (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2
Catheter Site Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Legionella Infection (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 2
Osteomyelitis (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 10 | 18
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pneumonia Legionella (Infections and infestations) | 0 | 1
Post Procedural Infection (Infections and infestations) | 1 | 0
Prostate Infection (Infections and infestations) | 0 | 1
Pseudomembranous Colitis (Infections and infestations) | 1 | 0
Pulmonary Mycosis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 4
Renal Abscess (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 7 | 5
Septic Shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 12
Urosepsis (Infections and infestations) | 2 | 2
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 8
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 3
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 2
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 2
Oxygen Saturation Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 3 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered State of Consciousness (Nervous system disorders) | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 2 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 4 | 2
Cognitive Disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Embolic Cerebral Infarction (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 2 | 1
Loss of Consciousness (Nervous system disorders) | 1 | 0
Nervous System Disorder (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Spinal Cord Compression (Nervous system disorders) | 3 | 5
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 6
Transient Ischaemic Attack (Nervous system disorders) | 1 | 3
Device Occlusion (Product Issues) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 7 | 6
Bladder Obstruction (Renal and urinary disorders) | 0 | 1
Calculus Bladder (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 13 | 6
Hydronephrosis (Renal and urinary disorders) | 0 | 4
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 3
Urinary Retention (Renal and urinary disorders) | 3 | 3
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 4
Testicular Pain (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 | 0
Coronary Angioplasty (Surgical and medical procedures) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 2 | 2
Aortic Dissection (Vascular disorders) | 0 | 1
Aortic Stenosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 4 | 1
Embolism (Vascular disorders) | 2 | 0
Haemodynamic Instability (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Hypertensive Urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Pelvic Venous Thrombosis (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+ Abiraterone Acetate - Prednisolone (N=489) | Apalutamide + Abiraterone Acetate - Prednisolone (N=490)
Anaemia (Blood and lymphatic system disorders) | 77 | 70
Hypothyroidism (Endocrine disorders) | 8 | 27
Abdominal Pain (Gastrointestinal disorders) | 25 | 24
Constipation (Gastrointestinal disorders) | 94 | 96
Diarrhoea (Gastrointestinal disorders) | 73 | 91
Dyspepsia (Gastrointestinal disorders) | 21 | 28
Nausea (Gastrointestinal disorders) | 76 | 84
Vomiting (Gastrointestinal disorders) | 35 | 39
Asthenia (General disorders) | 63 | 65
Fatigue (General disorders) | 134 | 164
Oedema Peripheral (General disorders) | 72 | 77
Pyrexia (General disorders) | 36 | 36
Influenza (Infections and infestations) | 28 | 20
Nasopharyngitis (Infections and infestations) | 57 | 52
Upper Respiratory Tract Infection (Infections and infestations) | 40 | 42
Urinary Tract Infection (Infections and infestations) | 49 | 37
Contusion (Injury, poisoning and procedural complications) | 49 | 34
Fall (Injury, poisoning and procedural complications) | 92 | 106
Rib Fracture (Injury, poisoning and procedural complications) | 23 | 25
Alanine Aminotransferase Increased (Investigations) | 57 | 20
Aspartate Aminotransferase Increased (Investigations) | 53 | 21
Blood Alkaline Phosphatase Increased (Investigations) | 34 | 19
Blood Pressure Increased (Investigations) | 17 | 26
Weight Decreased (Investigations) | 84 | 136
Weight Increased (Investigations) | 28 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 60 | 72
Hypercholesterolaemia (Metabolism and nutrition disorders) | 18 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 37 | 29
Hypokalaemia (Metabolism and nutrition disorders) | 73 | 79
Arthralgia (Musculoskeletal and connective tissue disorders) | 121 | 127
Back Pain (Musculoskeletal and connective tissue disorders) | 133 | 154
Bone Pain (Musculoskeletal and connective tissue disorders) | 48 | 34
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 45 | 30
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 50 | 48
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 46 | 50
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 27
Neck Pain (Musculoskeletal and connective tissue disorders) | 13 | 26
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 57 | 79
Dizziness (Nervous system disorders) | 46 | 61
Dysgeusia (Nervous system disorders) | 12 | 33
Headache (Nervous system disorders) | 63 | 79
Anxiety (Psychiatric disorders) | 16 | 28
Insomnia (Psychiatric disorders) | 30 | 46
Haematuria (Renal and urinary disorders) | 40 | 42
Pollakiuria (Renal and urinary disorders) | 31 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 43 | 41
Rash (Skin and subcutaneous tissue disorders) | 24 | 44
Hot Flush (Vascular disorders) | 56 | 74
Hypertension (Vascular disorders) | 122 | 144

LIMITATIONS AND CAVEATS:
This study used an electronic handheld device to collect responses for patient-reported outcome (PRO) questionnaires, which might have resulted in a lower-than-expected compliance due to unfamiliarity of the elderly population with the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT02257736/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02257736/SAP_001.pdf